CLINICAL TRIAL: NCT03089710
Title: The Effectiveness of Mini-fluid Challenge in Predicting Fluid Responsiveness During Prone Position Spine Surgery
Brief Title: Mini-fluid Challenge in Predicting Fluid Responsiveness During Prone Position Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201612021RIND
Record Dates: First submitted 2017-02-22; First posted 2017-03-24 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2018-10

CONDITIONS: Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mini-Fluid Challenge arm (Experimental): Fluid challenge test will be presented after induction of anesthesia at a steady state. Fluid challenge test includes 2 components: 100 ml colloid infusion in 1 min followed by 400 ml colloid infusion in 14 mins. Hemodynamic parameter after 1 minute of the end of the 1st and 2nd colloid infusion bolus will be collected.
  Applied colloid: hydroxyethyl starch
  Interventions: Other: Mini-fluid challenge

INTERVENTIONS:
Other: Mini-fluid challenge — Mini-fluid challenge test with 100mL colloid infusion in 1 min

SUMMARY:
Perioperative fluid management is crucial for patients' outcome. Muller et al developed a "Mini-fluid challenge method " to predict fluid responsiveness and the efficacy. The investigators design the study to investigate the effectiveness of mini-fluid challenge test in prone position surgery.

DETAILED DESCRIPTION:
Perioperative fluid management is crucial for patients' outcome. Series of studies have indicated that adequate fluid management optimizes the cardiac out put, improves tissue perfusion, thus decrease the risk of postoperative morbidity. Muller et al developed a "Mini-fluid challenge method " to predict fluid responsiveness and the efficacy. To the best of our knowledge, the efficacy of the test was not discussed in the perioperative care in prone position surgery. The investigators design the study to investigate the effectiveness of mini-fluid challenge test in prone position surgery.

ELIGIBILITY:
Inclusion Criteria: meet both of

1. Patients receiving scheduled prone position spine surgery
2. BMI 18.5~30 kg.m-2

Exclusion Criteria:

1. age younger then 20 yrs or elder than 80 yrs
2. pregnant women
3. patients in intensive care units
4. patients with the underlying disease including respiratory failure(FEV1/FVC < 70 % and FEV1 < 50%), heart failure(NYHA score =III、IV), kidney failure(eGFR< 60 ml.min-1.1.73m-2), liver failure
5. patients with ongoing infection
6. patients allergic to voluven

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Change of cardiac index after fluid loading | 3hr
  interpretate the correlation of mini-fluid challenge and conventional fluid challenge

SECONDARY OUTCOMES:
pulse pressure variation(PPV) | 3hr
  interpretate the correlation of PPV and conventional fluid challenge

OTHER OUTCOMES:
stroke volume variation(SVV) | 3hr
  interpretate the correlation of SVV and conventional fluid challenge
plethysmographic variation index(PVI) | 3hr
  interpretate the correlation of PVI and conventional fluid challenge

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided